CLINICAL TRIAL: NCT06659068
Title: Efficacy of Seluang Fish Oil (Rasbora Argyrotaenia) and Synbiotics Supplementation on CD4+CD25+ Foxp3+ T-regulator Cells, IL17/IL-10 Ratio, and Disease Activity in Systemic Lupus Erythematosus Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Yuniza, Principal investigator, Division of Allergy Immunology Faculty Member, Department of Internal Medicine, Universitas Sriwijaya/Mohammad Hoesin General Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4.3/D.XVIII.6.8/ETIK/208/2023
Record Dates: First submitted 2024-09-30; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Seluang fish oil; Rasbora argyrotaenia; Systemic Lupus Erythematosus; SLE; IL-17/IL-10 ratio; CD4+; CD25+; Foxp3+; T-regulator; Disease Activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: The study was designed as a single-center double-blind randomized controlled clinical trial. Participants were randomized into two groups receiving seluang fish oil and synbiotics supplementation, or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Seluang fish oil (Rasbora argyrotaenia) and Synbiotic (Experimental): Seluang fish oil (Rasbora argyrotaenia) and Synbiotic
  The patients were given a capsule containing seluang fish oil (Rasbora argyrotaenia) once a day and also synbiotic once a day
  Interventions: Dietary Supplement: Seluang fish oil (Rasbora argyrotaenia) and synbiotic
- Placebo (Placebo Comparator): Placebo
  The patients were given placebo capsules of seluang fish oil (Rasbora argyrotaenia) and synbiotics once a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Seluang fish oil (Rasbora argyrotaenia) and synbiotic — The patients received seluang fish oil (Rasbora argyrotaenia) and synbiotics (containing Lactobacillus helveticus R0052 60%, Bifidobacterium infantis R0033 20%, Bifidobacterium bifidum R0071 20% and frukto-oligosaccharide 80 mg) supplementation
  Arms: Seluang fish oil (Rasbora argyrotaenia) and Synbiotic
Dietary Supplement: Placebo — Patients received placebo capsules
  Arms: Placebo

SUMMARY:
The study aimed to evaluate the efficacy of seluang fish oil (Rasbora argyrotaenia) and synbiotics (containing Lactobacillus helveticus R0052 60%, Bifidobacterium infantis R0033 20%, Bifidobacterium bifidum R0071 20% and frukto-oligosaccharide 80 mg) supplementation compared to placebo towards Systemic Lupus Erythematosus disease activity Index (SLEDAI)-2K score, IL-17/IL-10 ratio and CD4+ CD25+ Foxp3+T-regulator levels in Systemic Lupus Erythematosus (SLE) patients. The current study was designed as a single-center double-blind randomized controlled clinical trial. The participants were voluntarily recruited 18-55 years old SLE patients diagnosed based on SLICC criteria, with mild to moderate disease activity, were clinically stable for ≥ 4 months (on prednison ≤ 20 mg/day or equivalent) and willingly ceased vitamin D and probiotic consumption during the trial study. Participants were randomized into two groups receiving seluang fish oil and synbiotics supplementation, or placebo. Evaluations were conducted on week 4, 8 and 12 for clinical symptoms, side effects and adherence. IL-17/IL-10 ratio and CD4+ CD25+ Foxp3+T-regulator levels were evaluated at the beginning and at the end of the 12 week trial for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the SLICC criteria
* Patients with mild to moderate SLE (mild if SLEDAI-2K score < 6 and moderate if SLEDAI-2K score: 6-12)
* Aged 18-55 years
* Willing to stop consuming vitamin D or multivitamin supplements containing vitamin D for at least 3 weeks before participating in the study
* Willing to stop consuming probiotics that were previously taken for at least 1 week before participating in the study
* If using prednisone, the dose must be stable (corticosteroid equivalent ≤ 20 mg/day) for at least 4 weeks before the study
* Willing to sign informed consent

Exclusion Criteria:

* Patients with severe SLE
* Patients with SLE with hypercalcemia (> 2.60 mmol/l)
* Patients with SLE with liver dysfunction: serum Aspartate Transferase (AST) - and Alanine Transferase (ALT) levels > 2 times the normal value or total serum bilirubin > 1.5 times the normal value
* Patients undergoing hemodialysis or patients with serum creatinine > 2.5 mg/dL
* Pregnant patients
* Patients with SLE with immunocompromised conditions such as HIV
* Patients with SLE with chronic infections such as pulmonary tuberculosis
* Patients currently undergoing antibiotic therapy

Drop out criteria:

* Patients who have been off medication for more than 3 weeks
* Patients who have passed away
* Patients who consume yogurt or supplements containing probiotics/synbiotics more than once consecutively in 1 week
* Patients who experience a change in immunosuppressive agents during the study
* Patients who are hospitalized due to a worsening condition during the intervention period
* Loss to follow-up

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
CD4+CD25+Foxp3+ regulatory T cells, | From enrollment to the end of the treatment at 12 weeks
  To determine the effectiveness of adding seluang fish oil extract capsules with synbiotics compared to placebo in CD4+CD25+Foxp3+ regulatory T cells concentration change
IL-17/IL-10 ratio | From enrollment to the end of the treatment at 12 weeks
  To determine the effectiveness of adding seluang fish oil extract capsules with synbiotics compared to placebo in IL-17/IL-10 ratio changes
SLEDAI-2K score | From enrollment to the end of the treatment at 12 weeks
  To determine the effectiveness of adding seluang fish oil extract capsules with synbiotics compared to placebo towards SLEDAI-2K score changes

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Hoesin General Hospital, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Partan RU, Hidayat R, Saputra N, Rahmayani F, Prapto H, Yudha TW. Seluang Fish (Rasbora Spp.) Oil Decreases Inflammatory Cytokines Via Increasing Vitamin D Level in Systemic Lupus Erythematosus. Open Access Maced J Med Sci. 2019 May 5;7(9):1418-1421. doi: 10.3889/oamjms.2019.308. eCollection 2019 May 15. PMID 31198446
- [Background] Widhani A, Djauzi S, Suyatna FD, Dewi BE. Changes in Gut Microbiota and Systemic Inflammation after Synbiotic Supplementation in Patients with Systemic Lupus Erythematosus: A Randomized, Double-Blind, Placebo-Controlled Trial. Cells. 2022 Oct 29;11(21):3419. doi: 10.3390/cells11213419. PMID 36359816
- [Background] Partan RU, Mart Salim E, Hidayat R. The potential role of seluang fish oil (Rasbora Spp) in improving calcium, zinc and vitamin d3 deficiencies. International Journal of Oceans and Oceanography. 2017: 11; 2. 285-29